CLINICAL TRIAL: NCT03254693
Title: STRATEGIES FOR BONDING TO ENAMEL USING A UNIVERSAL ADHESIVE ON SELF-ETCHING MODE
Brief Title: BONDING TO ENAMEL USING A UNIVERSAL ADHESIVE
Acronym: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Eloisa Andrade de Paula, Doctor, Universidade Estadual do Oeste do Paraná
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 56013116.0.0000.0107
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Clinical Trial
Keywords: Non-carious cervical lesions; Universal system; Longevity.

STUDY DESIGN:
Intervention Model Description: This was a double-blind, equivalence superiority, split-mouth randomized clinical trial. The restoration procedures were carried out within the clinics of the Dental School of the Federal University of Rio de Janeiro in Rio de Janeiro (Rio de Janeiro, Brazil) and at the State University Oeste do Paraná in Cascavel (Paraná, Brazil) from July 2016 to August 2017.
Who Masked: Participant, Outcomes Assessor
Masking Description: staff member not involved in the research protocol performed the randomization process with computer-generated tables. Details of the allocated groups were recorded on cards contained in sequentially numbered, opaque, sealed envelopes. Opening the envelope only on the day of the restorative procedure guaranteed the concealment of the random sequence. The examiners were not involved with the restoration procedures and therefore blinded to the group assignment, performed the clinical evaluation. Patient were also blinded to group assignment in a double-blind randomized clinical trial design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1-step self-etch approach (SE) (Active Comparator): According to the manufacturer's instructions.
  Interventions: Combination Product: 1-step self-etch approach (SE)
- selective enamel etching (SEE) (Active Comparator): According to the manufacturer's instructions.
  Interventions: Combination Product: selective enamel etching (SEE)
- 1-step self-etch for double time (SE2X) (Experimental): According to the manufacturer's instructions, but for the double time (20 s) in the each application.
  Interventions: Other: 1-step self-etch for double time (SE2X)
- 1-step self-etch additional layer (SE1+) (Experimental): According to the manufacturer's instructions, but apply tree times.
  Interventions: Other: 1-step self-etch additional layer (SE1+)

INTERVENTIONS:
Combination Product: 1-step self-etch approach (SE) — Application mode - Do not use etchan. According to the manufacturer's instructions.
  Other Names: SE
  Arms: 1-step self-etch approach (SE)
Combination Product: selective enamel etching (SEE) — Application mode - Etch only on enamel for 15 s. Rinse for 15s. Air dry to remove excess water.According to the manufacturer's instructions.
  Other Names: SEE
  Arms: selective enamel etching (SEE)
Other: 1-step self-etch for double time (SE2X) — Application mode - Do not use etchan. According to the manufacturer's instructions, but for the double time (20 s) in the each application.
  Other Names: SE2X
  Arms: 1-step self-etch for double time (SE2X)
Other: 1-step self-etch additional layer (SE1+) — Application mode - Do not use etchan. According to the manufacturer's instructions, but apply tree times.
  Other Names: SE1+
  Arms: 1-step self-etch additional layer (SE1+)

SUMMARY:
Objective: This double-blind randomized clinical trial evaluates strategies for improving the bonding of universal adhesive to enamel in non-carious cervical lesions (NCCL) of a new universal multi-mode adhesive (Ambar Universal; FGM).

Methods: A total of 134 restorations were randomly placed in 19 patients according to the following groups: SE - Self-etch; SEE - Selective etching; SE2X - Self-etch doble time; SE1+ - Self-etch additional layer. The resin composite Opallis (FGM) was placed incrementally. The restorations were evaluated after one week (baseline), 6 and 12 months, using the FDI and USPHS criteria. Statistical analyses were performed using appropriate tests (=0.05).

DETAILED DESCRIPTION:
Interventions: restorative procedure All the patients selected for this study received dental prophylaxis with a suspension of pumice and water in a rubber cup and signed an informed consent form two weeks before the restorative procedures.

The degree of sclerotic dentin from the NCCLs was measured according to the criteria described by Swift and others. The cavity dimensions in millimeters (height, width, and depth), the geometry of the cavity (evaluated by profile photograph and labeled at <45o, 45o-90o, 90o<135o, and >135o), the presence of an antagonist, and the presence of attrition facets were observed and recorded. Pre-operative sensitivity was also evaluated by applying air for 10 s from a dental syringe placed 2 cm from the tooth surface and with an explorer. These features were recorded to allow comparison of the baseline features of the dentin cavities among experimental groups.

To calibrate the restorative procedure, the study director placed one restoration of each group to identify all steps involved in the application technique. Then, the two operators, who were resident dentists with more than five years of clinical experience in operative dentistry, placed four restorations, one of each group, under the supervision of the study director in a clinical setting. The restoration failures were shown to the operators prior to starting the study. At this point, the operators were considered calibrated to perform the restorative procedures.

The operators restored all teeth. All participants received four restorations, one of each experimental group in different lesions previously selected according to the inclusion criteria.

Before restorative procedures, the operators anesthetized the teeth with a 3% mepivacaine solution (Mepisv, Nova DFL, Rio de Janeiro, RJ, Brazil) and cleaned all lesions with pumice and water in a rubber cup, followed by rinsing and drying. Then, shade selection was made using a shade guide.

Cleaning of all lesions with pumice and water in a rubber cup was carried out, followed by rinsing and drying. Using a shade-selection guide, the proper shade of the composite was determined. Following the ADA guidelines, the operators did not prepare any additional retention or bevel.

The NCCLs received the multimode adhesive system applied in different modes: 1-step self-etch approach (SE), selective enamel etching (SEE), 1-step self-etch applied for double time in the enamel (SE2X), 1-step self-etch approach with additional layer (SE1+) was applied as described below. The compositions, more details regarding the adhesion strategies used and batch numbers are described in Table 2.

The adhesives were light-cured with a LED light-curing unit (1,000 mW/cm2) (Radii-cal), according to the manufacturer's instructions (Table 2). Opallis (FGM) composite resin was used in 2 to 3 increments, each one being light-cured (Radii-cal) for 30 s. The restorations were finished immediately with fine #2200 diamond burs (KG Sorensen). Polishing was performed with rubber points (Astropol, Ivoclar Vivadent, Liechtenstein).

ELIGIBILITY:
Inclusion Criteria:

* Participants had to be in good general health.
* At least 18 years old
* Have an acceptable oral hygiene level
* Present at least 20 teeth under occlusion
* At least four NCCLs in four different teeth
* These lesions had to be non-carious, non-retentive, deeper than 1 mm, and involve both the enamel and dentin of vital teeth without mobility.
* The cavo-surface margin could not involve more than 50% of enamel, and all lesions had cervical margins ending in dentin.

Exclusion Criteria:

* Participants had not be in good general health.
* At less 18 years old
* Have not an acceptable oral hygiene level
* Present at less 20 teeth under occlusion
* At less four NCCLs in four different teeth, these lesions had not be non-carious, retentive and involve only enamel of vital teeth with mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Retention | 6 montths
  The primary clinical endpoint was restoration retention/fracture.

SECONDARY OUTCOMES:
Marginal Adaptation | 6 months
  Restoration marginal adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Scheffer, Master, Study Chair — Universidade Estadual do Oeste do Paraná
Locations (1):
- Universidade Estadual do Oeste do Paraná, Cascavel, Paraná, Brazil